CLINICAL TRIAL: NCT05800093
Title: Proteomics and Genomics Combined With CT to Predict CVD
Acronym: PREDICT-CVD
Status: Active, not recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL81913.018.22
Record Dates: First submitted 2023-03-13; First posted 2023-04-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates plaque progression and characteristics in patients with coronary atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 50 and 75 years old
* Subjects at intermediate to high risk for ASCVD
* Asymptomatic patients without cardiac chest pain
* Evidence of atherosclerosis on baseline CCTA

Exclusion Criteria:

* Renal insufficiency, defined as eGFR < 30 ml/min
* History of cardiovascular events (myocardial infarction, peripheral artery disease and ischemic stroke)
* Use of lipid lowering therapy other than statin, ezetimibe or bempedoic acid monotherapy
* Change in lipid lowering therapy in the last 6 months
* Use of more than two antihypertensive agents
* No coronary atherosclerosis at baseline imaging
* Active malignancy requiring treatment
* Atrial fibrillation
* Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients between 50 and 75 years old with nonobstructive coronary artery disease
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Coronary Artery Disease Progression | Through study completion, between 130-156 weeks

SECONDARY OUTCOMES:
Presence of obstructive stenosis | Through study completion, between 130-156 weeks
Progression in number of significant (>50%) and severe (>70%) stenoses | Through study completion, between 130-156 weeks
Total plaque volume progression | Through study completion, between 130-156 weeks
Calcified plaque volume progression | Through study completion, between 130-156 weeks
Non-calcified plaque volume progression | Through study completion, between 130-156 weeks
Low-attenuation plaque volume progression | Through study completion, between 130-156 weeks
Change in Pericoronary Adipose Tissue CT-Attenuation | Through study completion, between 130-156 weeks
CAD-RADS progression (yes/no) | Through study completion, between 130-156 weeks
Progression in number of high-risk plaque characteristics (yes/no) | Through study completion, between 130-156 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik SG Stroes, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No